CLINICAL TRIAL: NCT04666948
Title: A Multicentric, Randomised Controlled Clinical Trial to Study the Impact of Bedside Model-informed Precision Dosing of Vancomycin in Critically Ill Children
Brief Title: Precision Dosing of Vancomycin in Critically Ill Children
Acronym: BENEFICIAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Belgium Health Care Knowledge Centre (Other Government); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-5429
Record Dates: First submitted 2020-11-28; First posted 2020-12-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Vancomycin
Keywords: vancomycin; model-informed precision dosing; critically ill children; dose calculator
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and parents or legal representatives are blinded for the allocation to the intervention or standard-of-care arm until the end of study.
  the statistician is kept blinded until after data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Vancomycin treatment (Active Comparator): Vancomycin standard-of-care dosing and therapeutic drug monitoring, according to institutional guidelines during 30 day study period
  Interventions: Drug: Vancomycin
- vancomycin model-informed precision dosing (Experimental): Area Under the Concentration (AUC)-time curve/MIC-based model-informed precision dosing of vancomycin using a CE labelled dosing calculator during 30 day study period
  Interventions: Device: vancomycin model-informed precision dosing; Drug: Vancomycin

INTERVENTIONS:
Device: vancomycin model-informed precision dosing — A CE labelled dosing calculator is used for a priori and a posteriori calculation of vancomycin dose using a target AUC between 400-600 mg*h/L
  Other Names: dosing calculator
  Arms: vancomycin model-informed precision dosing
Drug: Vancomycin — Vancomycin treatment

SUMMARY:
The overall objective of this project is to investigate the large-scale utility of MIPD of vancomycin at point-of-care in ICU children. This evaluation includes a comparison with the more standard approach on Clinical and patient-oriented measures.

DETAILED DESCRIPTION:
Vancomycin is an antibiotic with a narrow therapeutic-toxic margin. This means that the minimum and maximum target blood target levels differ little from each other. Too low concentrations will reduce the effect of the antibiotic; higher concentrations may result in serious side effects, including renal toxicity. Vancomycin dosing tailored to the critically ill child is challenging.

Currently, the starting dose of vancomycin is calculated on a milligram per kilogram basis, which is the same for all patients. The dose is then adjusted based on a measured vancomycin blood concentration (if too high or too low). Despite this measurement, quickly achieving target concentrations remains a major challenge.

This multicenter, individual randomized study investigates the added value of a user-friendly computer program for calculating the vancomycin dose in critically ill children, compared to the current standard-of-care. Specifically, the investigators will study whether the use of this computer program leads to a shorter time to reach target concentrations, a reduction in the number and severity of side effects on the kidney, a reduction in patient burden, and a reduction in time to cure and duration of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* age: 0-18 years
* admitted to ICU or PHO unit
* suspected or confirmed Gram positive infection
* planned to start on intravenous intermittent or continuous infusion vancomycin treatment
* informed consent signed by parents or legal representatives
* not previously enrolled in this trial

Exclusion Criteria:

* extracorporeal treatment at inclusion or started during treatment (extracorporeal membrane oxygenation, dialysis, body cooling)
* n or p RIFLE category failure at inclusion (Day 0) (see section 8.1.2. screening)
* Known chronic kidney disease as defined by the KDIGO definition as: structural or functional abnormalities of the kidney regardless of GFR for < 3 months or GFR < 60ml/min/1.73m² for ≥ 3 months. eGFR is estimated using the modified Schwartz equation
* patient death is deemed imminent and inevitable

Ages: 0 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 314 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reaching target 24hAUC/MIC | 24 to 48 hours after start vancomycin treatment
  therapeutic AUC/MIC target range is 400-600

SECONDARY OUTCOMES:
Proportion of patients with (worsening) acute kidney injury during vancomycin treatment | from start date of vancomycin treatment until stop date vancomycin treatment or study day 30, whichever comes first
  AKI categories are defined according to the neonatal and pediatric RIFLE criteria
Proportion of patients reaching target 24h AUC/MIC | 48-72 hours after start vancomycin treatment
  therapeutic AUC/MIC target range is 400-600
Time to clinical cure | 30 day study period
  Time to clinical cure is defined as the time interval (in days) from start to completion of the vancomycin vancomycin treatment, without recommencement of antibiotics for the same indication within 48h after stop.
Ward unit length-of-stay | 30 day study period
  Ward unit length-of-stay is calculated from day of ward unit admission to day of ward unit discharge.
Hospital length-of-stay | 30 day study period
  Hospital unit length-of-stay is calculated from day of hospital admission to day of hospital discharge.
30 day all cause mortality | 30 day study period
  30 day all cause mortality is measured 30 days after randomisation.

OTHER OUTCOMES:
Cumulative number of additional blood samples during treatment in patients with clinical cure | from start date of vancomycin treatment until stop date vancomycin treatment or study day 30, whichever comes first in patients with clinical cure
  An additional blood sample is defined as a sample for vancomycin TDM taken at another timepoint of routine biochemical monitoring samples.
Number of additional blood samples to first target attainment during vancomycin treatment | from start date of vancomycin treatment until date of first vancomycin target attainment or study day 30, whichever comes first
  An additional blood sample is defined as a sample for vancomycin TDM taken at another timepoint of routine biochemical monitoring samples.
Proportion of patients reaching target 24h AUC/MIC | 72-96 hours after start vancomycin treatment
  therapeutic AUC/MIC target range is 400-600
Number of dose adjustments to first target attainment | from start date vancomycin treatment until date of first vancomycin target attainment or study day 30, whichever comes first
  Target in Model-Informed Precision Dosing arm: 24h AUC/MIC : 400-600; in comparator arm: target concentration range according to institutional guidelines
Number of trough sampling time errors | from start date of vancomycin treatment until stop date vancomycin treatment or study day 30, whichever comes first
  only measured for intermittent dosing regimens in the comparator arm.
Cumulative vancomycin dose and AUC | from start date of vancomycin treatment until stop date vancomycin treatment or study day 30, whichever comes first
  Total cumulative dose and exposure (AUC) during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pieter De Cock, Prof, Principal Investigator — University Hospital, Ghent
Locations (7):
- Belgium (7):
  - Erasme, Brussels, Brussels Capital
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - Cliniques universitaires de Saint Luc, Brussels
  - Hopital universitaire de Reine Fabiola, Brussels
  - UZ Brussel, Brussels
  - Ghent University Hospital, Ghent
  - UZ Leuven, Leuven